CLINICAL TRIAL: NCT04342403
Title: Clinical Studies Network Research Trial: Development of an On-Line Sarcoidosis Assessment Platform (OSAP) to Validate Sarcoidosis Phenotypes and Monitor Disease Burden Longitudinally
Brief Title: Patient Reported Outcome Instruments in Sarcoidosis
Acronym: OSAP-PRO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Cincinnati (Other)
Collaborators: Foundation for Sarcoidosis Research (Other); Albany Medical College (Other)
Responsible Party: Principal Investigator, Robert P Baughman, Professor, University of Cincinnati
Other Study IDs: 2015-7046
Record Dates: First submitted 2020-04-08; First posted 2020-04-13 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Sarcoidosis
MeSH Terms: conditions — Sarcoidosis | interventions — Respiratory Function Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sarcoidosis: Patients with sarcoidosis willing to participate
  Interventions: Diagnostic Test: Quality of Life

INTERVENTIONS:
Diagnostic Test: Quality of Life — Quality of life instruments including King's Sarcoidosis Questionnaire (KSQ) and Sarcoidosis Assessment Tool (SAT)
  Other Names: Pulmonary function testing

SUMMARY:
Evaluate change of quality of life of sarcoiodosis patients over a six months using various quality of life instruments including a monthly smart phone app.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of sarcoidosis by established criteria.
* Patient has completed pulmonary function tests (spirometry) as per standard of care at the enrollment visit.
* Ability to understand and read English at least at a 7th grade level.
* Have access to a computer, iPad, smart phone, or another electronic device that will support the on-line sarcoidosis assessment platform.
* The subject is willing to wear a daily activity and sleep tracker wristband (Fitbit ™ wristband) for 6 months.

Exclusion Criteria:

• Life expectancy of < 1 year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients followed at sarcoidosis clinics across United States
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
KSQ | 6 months
  Change in KSQ

SECONDARY OUTCOMES:
SAT | 6 Months
  Change in SAT
Visual Analog Scale (VAS) | 6 Months
  Change in VAS
Forced Vital Capacity (FVC) | 6 months
  Change in FVC percent predicted

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Albany Medical Center, Albany, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No
none at this time

REFERENCES:
- [Derived] Judson MA, Yucel R, Preston S, Chen ES, Culver DA, Hamzeh N, Lower EE, Sweiss NJ, Valeyre D, Veltkamp M, Victorson DE, Beaumont JL, Singh N, Shivas T, Vancavage R, Baughman RP. The association of baseline sarcoidosis measurements with 6-month outcomes that are of interest to patients: Results from the On-line Sarcoidosis Assessment Platform Study (OSAP). Respir Med. 2022 May;196:106819. doi: 10.1016/j.rmed.2022.106819. Epub 2022 Mar 18. PMID 35358810